CLINICAL TRIAL: NCT00101933
Title: SANTE - Stimulation of the Anterior Nucleus of the Thalamus for Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1604
Record Dates: First submitted 2005-01-18; First posted 2005-01-19 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Epilepsy
Keywords: Deep brain stimulation, DBS, SANTE
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active Stimulation
  Interventions: Device: Medtronic DBS Therapy for epilepsy
- 2 (Sham Comparator): No Stimulation
  Interventions: Device: Medtronic DBS Therapy for epilepsy

INTERVENTIONS:
Device: Medtronic DBS Therapy for epilepsy — Stimulation On
  Arms: 1
Device: Medtronic DBS Therapy for epilepsy — Stimulation Off
  Arms: 2

SUMMARY:
The purpose of this research is to study the safety and effectiveness of bilateral stimulation of the anterior nucleus of the thalamus as adjunctive therapy for reducing the frequency of seizures in adults diagnosed with epilepsy characterized by partial-onset seizures, with or without secondary generalization, that are refractory to antiepileptic medications.

DETAILED DESCRIPTION:
Medtronic, Inc. is sponsoring an investigational study of the Medtronic DBS Therapy for epilepsy, the company's deep brain stimulation (DBS) therapy for patients with refractory epilepsy. Epilepsy is a condition that affects 2.3 million Americans, and about one-third of these patients are refractory, or continue to experience seizures despite a wide range of treatment options.

The prospective, randomized, double-blind trial uses existing technology to test whether bilateral stimulation of the anterior nucleus of the thalamus can safely and effectively reduce seizure frequency in patients with epilepsy. It includes enrollment of 157 patients at 17 sites in the U.S. 110 patients were implanted and monitored for 13 months following implant, with long-term follow-up until the device is approved or the study is stopped. 109 of the 110 implanted subjects were randomized to Active stimulation or Control.

Patients in the active group, who received neurostimulation, were monitored for a reduction in seizure rates compared to the control group, who did not receive neurostimulation during the three-month double-blind phase. After the double-blind phase, all patients received neurostimulation.

Candidates for the trial were adults with partial-onset epilepsy for whom at least three antiepileptic drugs have proven ineffective. They were to have had an average of six or more seizures per month. Candidates continued to receive their epilepsy medications while participating in the trial.

Deep brain stimulation therapy has already received approval in the United States, Europe, Canada, and Australia for the treatment of Essential Tremor and Parkinson's disease. Deep brain stimulation is not approved in the United States for the treatment of epilepsy.

ELIGIBILITY:
Relevant Inclusion and Exclusion Criteria are listed below.

Inclusion Criteria

* Partial-onset seizures with or without secondary generalization. The final determination shall be made by the Investigator based on a clinical description of the seizures and previous diagnostic testing that includes, at a minimum, video/clinical EEG that captured at least one ictal event.
* Anticipated average of 6 or more partial-onset seizures (with or without secondary generalized seizures) per month during the Baseline Phase, with no more than 30 days between seizures during the Baseline Phase.
* Refractory to antiepileptic drugs (AEDs). Patients will be considered refractory if they have failed at least three AEDs due to lack of efficacy.
* Receiving one to four currently marketed AEDs
* Be between 18 and 65 years of age at the time of lead implant

Exclusion Criteria:

* Multilobar (>3 different lobes) anatomic areas of seizure onset
* Symptomatic generalized epilepsy
* Previous diagnosis of psychogenic/non-epileptic seizures
* Presence of implanted electrical stimulation medical device anywhere in the body (e.g., cardiac pacemakers, spinal cord stimulator) or any metallic implants in the head (e.g., aneurysm clip, cochlear implant). Vagal nerve stimulators are allowed if the device has been turned off for at least 30 days prior to the Baseline Week -12 visit and the patient agrees to have the generator explanted prior to or at the time of the Kinetra Neurostimulator implant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2003-12 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2017-10 (Actual)

REFERENCES:
- [Background] Miller PM, Gross RE. Wire tethering or 'bowstringing' as a long-term hardware-related complication of deep brain stimulation. Stereotact Funct Neurosurg. 2009;87(6):353-9. doi: 10.1159/000236369. Epub 2009 Sep 10. PMID 19752594
- [Result] Fisher R, Salanova V, Witt T, Worth R, Henry T, Gross R, Oommen K, Osorio I, Nazzaro J, Labar D, Kaplitt M, Sperling M, Sandok E, Neal J, Handforth A, Stern J, DeSalles A, Chung S, Shetter A, Bergen D, Bakay R, Henderson J, French J, Baltuch G, Rosenfeld W, Youkilis A, Marks W, Garcia P, Barbaro N, Fountain N, Bazil C, Goodman R, McKhann G, Babu Krishnamurthy K, Papavassiliou S, Epstein C, Pollard J, Tonder L, Grebin J, Coffey R, Graves N; SANTE Study Group. Electrical stimulation of the anterior nucleus of thalamus for treatment of refractory epilepsy. Epilepsia. 2010 May;51(5):899-908. doi: 10.1111/j.1528-1167.2010.02536.x. Epub 2010 Mar 17. PMID 20331461
- [Result] Troster AI, Meador KJ, Irwin CP, Fisher RS; SANTE Study Group. Memory and mood outcomes after anterior thalamic stimulation for refractory partial epilepsy. Seizure. 2017 Feb;45:133-141. doi: 10.1016/j.seizure.2016.12.014. Epub 2016 Dec 23. PMID 28061418
- [Result] Salanova V, Witt T, Worth R, Henry TR, Gross RE, Nazzaro JM, Labar D, Sperling MR, Sharan A, Sandok E, Handforth A, Stern JM, Chung S, Henderson JM, French J, Baltuch G, Rosenfeld WE, Garcia P, Barbaro NM, Fountain NB, Elias WJ, Goodman RR, Pollard JR, Troster AI, Irwin CP, Lambrecht K, Graves N, Fisher R; SANTE Study Group. Long-term efficacy and safety of thalamic stimulation for drug-resistant partial epilepsy. Neurology. 2015 Mar 10;84(10):1017-25. doi: 10.1212/WNL.0000000000001334. Epub 2015 Feb 6. PMID 25663221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 157 subjects were enrolled in the study from 11 DEC 2003 through 23 FEB 2007 from 17 centers in US.
Pre-assignment Details: 47 of 157 subjects exited prior to implant due to not meeting in/exclusion criteria, withdrawal of consent to participate, etc. Of the remaining 110 subjects, 109 subjects were randomized. Those 109 subjects were used for objectives between randomization groups while all 110 implanted subjects were used for long term safety objectives.
Groups:
- Active Stimulation: This group contains subjects who were implanted and randomized to receive active stimulation during the blinded phase of the study.
- No Stimulation: This group contains subjects who were implanted and randomized to receive no stimulation during the blinded phase of the study.
Period: Overall Study
Arm/Group | Active Stimulation | No Stimulation
Started | 54 | 55
Completed | 54 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation | No Stimulation | Total
Number analyzed (Participants) | 54 | 55 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 55 | 109
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (11.1) | 36.8 (11.5) | 36.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 25 | 30 | 55
Region of Enrollment [Number; unit: participants]
  United States | 54 | 55 | 109

OUTCOME MEASURES:

1. Primary Outcome: Primary Analysis: Change in Seizure Rate
Description: A protocol-prespecified generalized estimating equations (GEE) analysis was used to evaluate the treatment effect on seizure frequency. The final GEE model for the primary objective evaluation included treatment effect, log of the baseline seizure count, log of age, visit (categorical), treatment-by-visit interaction (categorical), and the offset (the number of days the diary was recorded in each month).
Time Frame: Through the end of the three-month blinded phase
Population: This analysis used the protocol-prespecified "Primary analysis data set" which required that subjects had at least 70 days of diary in the blinded phase. One control subject was not included in this analysis as they had 66 of the required 70 days.
Measure: Median (Inter-Quartile Range); unit: Percentage change from baseline
Arm/Group | Active Stimulation | No Stimulation
Number analyzed (Participants) | 54 | 54
Percentage change from baseline | -40.4 [-62.9 to -21.6] | -14.5 [-50.3 to 20.0]
Statistical Analysis 1: Comparison: Active Stimulation vs No Stimulation; The numbers presented are the percentage reduction in the number of seizures in each group. A negative percentage change indicates a seizure reduction; Test type: Superiority or Other; p = 0.0017, Generalized Estimating Equations — Since a treatment-by-visit interaction remains in the final model, the results were analyzed by visit. The results shown are for the last month in the blinded phase (month 3-4); This analysis is adjusted for significant baseline covariates

2. Secondary Outcome: Adverse Events Experienced With the Medtronic DBS System
Description: The results are for the follow-up after device implantation through Year 2 and summarized are events that occurred in greater than 5% of subjects. Only events related to the device, therapy, or surgery are included. These abbreviations were used:
  * General dis...=General disorders and administration site conditions
  * Injury, poison...=Injury, poisoning and procedural complications
  * Ther.=Therapeutic.
  For this summary, adverse events are reported as 'MedDRA System Organ Class - adverse event'.
Time Frame: Through Year 2 of the long-term follow-up phase
Population: This analysis used all subjects who were implanted and received stimulation. One subject was implanted but was not subsequently randomized, but did receive stimulation. This subject has been included for the purposes of this analysis for a total of 110 subjects, as opposed to the 109 stated in the participant flow.
Measure: Number; unit: participants
Groups:
- All Implanted Subjects: This group contains all subjects who were implanted. This includes one additional subject over those that were randomized.
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 110
participants
  Total # of participants at risk | 110
  Infections and infestations-Implant site infection | 10
  Nervous system disorders-Paresthesia | 23
  Nervous system disorders-Sensory disturbance | 8
  Nervous system disorders-Dizziness | 6
  Nervous system disorders-Memory impairment | 7
  General dis...-Implant site pain | 18
  General dis...-Discomfort | 8
  General dis...-Lead(s) not within target | 9
  General dis...-Implant site inflammation | 6
  Injury, poison...-Post procedural pain | 7

3. Secondary Outcome: Incidence of Sudden Unexplained Death in Epilepsy (SUDEP)
Description: The number presented is for Definite and Probable SUDEP. The rate is calculated per 1000 subject years of follow-up. The confidence interval is the 95% Poisson confidence interval. Per protocol, only definite and probable SUDEP classifications were included in the calculation.
  The results shown are for the entire study follow-up after device implantation.
Time Frame: Inclusive of all study follow-up after device implantation (mean follow-up 3.7 years)
Population: This analysis used all subjects who were implanted and received stimulation. One subject was implanted but was not subsequently randomized, but did receive stimulation. This subject has been included for the purposes of this analysis for a total of 110 subjects included in this analysis.
Measure: Number; unit: Number of subjects experiencing SUDEP
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 110
Number of subjects experiencing SUDEP | 2 [0.60 to 17.79]
Statistical Analysis 1: Comparison: All Implanted Subjects; Test type: Superiority or Other; No statistical test; Rate per 1000 years of stimulation = 4.9, 95% CI 2-sided [0.60 to 17.79] — The rate is calculated per 1000 subject years of follow-up based on 406 subject years of stimulation. The confidence interval is the 95% Poisson confidence interval. Per protocol, only definite and probable SUDEP were included in the calculation

4. Secondary Outcome: Seizure Responder Rate
Description: A responder is defined as a subject with greater than or equal to 50% reduction in seizures as compared with baseline.
Time Frame: Through the end of the three-month blinded phase
Population: This analysis used the "Primary analysis data set" which required that subjects had at least 70 days of diary in the blinded phase. One control subject was not included in this analysis as they had 66 of the required 70 days.
Measure: Number; unit: Number of participants
Arm/Group | Active Stimulation | No Stimulation
Number analyzed (Participants) | 54 | 54
Number of participants | 16 | 14
Statistical Analysis 1: Comparison: Active Stimulation vs No Stimulation; Fisher's Exact test. The numbers presented in this analysis are the number of subjects who were responders based on a responder definition including all subjects with 50% or greater improvement in total seizure count; Test type: Superiority or Other; p = 0.830, Fisher Exact

5. Secondary Outcome: Change in Percentage of Days Seizure-free
Description: Difference between active group and control group in percentage change in seizure-free days over the entire blinded phase as compared to the entire baseline phase. The number of seizure-free days was normalized to 84-day baseline and blinded phases for each subject.
Time Frame: Through the end of the three-month blinded phase
Population: This analysis used the "Primary analysis data set" which required that subjects had at least 70 days of diary in the blinded phase. In addition, percentage change was not calculated for subjects who had no seizure-free days during the baseline phase.
Measure: Median (Inter-Quartile Range); unit: Percentage change from baseline
Arm/Group | Active Stimulation | No Stimulation
Number analyzed (Participants) | 50 | 50
Percentage change from baseline | 15.3 [7.6 to 38.3] | 8.8 [-0.5 to 26.5]
Statistical Analysis 1: Comparison: Active Stimulation vs No Stimulation; Test type: Superiority or Other; p = 0.105, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percentage Change in the Maximum Length of Seizure-free Intervals
Description: Difference between active group and control group in percentage change in the maximum length of seizure-free intervals over the entire blinded phase as compared to the entire baseline phase.
Time Frame: Through the end of the three-month blinded phase
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Percentage change from baseline
Arm/Group | Active Stimulation | No Stimulation
Number analyzed (Participants) | 54 | 54
Percentage change from baseline | 35.0 [0 to 129] | 24.0 [0 to 100]
Statistical Analysis 1: Comparison: Active Stimulation vs No Stimulation; Test type: Superiority or Other; p = 0.498, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Proportion of Treatment Failures
Description: A treatment failure was defined in the protocol as a subject who 1) required 3 or more doses of rescue medication within 48 hours, 3 times during the blinded phase; or 2) had 3 episodes of convulsive status epilepticus during the blinded phase.
Time Frame: Through the end of the three-month blinded phase
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Active Stimulation | No Stimulation
Number analyzed (Participants) | 54 | 54
participants | 0 | 0
Statistical Analysis 1: Comparison: Active Stimulation vs No Stimulation; Test type: Superiority or Other; p = 1.0, Fisher Exact

8. Primary Outcome: Alternative Primary Analysis: Change in Seizure Rate
Description: A generalized estimating equations (GEE) analysis was used to evaluate the treatment effect on seizure frequency. With one outlier subject removed, the GEE model for this alternative analysis included treatment effect, log of the baseline seizure count, log of age, visit (categorical), and the offset (the number of days the diary was recorded in each month).
Time Frame: Through the end of the three-month blinded phase
Population: This analysis used the protocol-prespecified "Primary analysis data set" with one additional outlier subject removed from the active group. This subject had 210 stimulation initiated seizures within 48 hours of the device being turned on and was determined to be an outlier using both a statistical and clinical rationale.
Measure: Median (Inter-Quartile Range); unit: Percentage change from baseline
Arm/Group | Active Stimulation | No Stimulation
Number analyzed (Participants) | 53 | 54
Percentage change from baseline | -35.0 [-53.9 to -14.5] | -21.1 [-51.5 to 7.5]
Statistical Analysis 1: Comparison: Active Stimulation vs No Stimulation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0387, Generalized Estimating Equations — Since a visit-by-treatment interaction did not remain in the final model, the results shown are for the entire blinded phase; This analysis is adjusted for significant baseline covariates

9. Other Pre Specified Outcome: Change in Most Severe Seizures
Description: Seizures were recorded on daily seizure diaries. The subject recorded the number of seizures by seizure type on the seizure diary. The subject also noted at baseline, of those they had ever experienced, which seizure they considered to be "most severe."
Time Frame: Through the end of the three-month blinded phase
Population: This analysis used the "Primary analysis data set". In addition, the protocol prespecified that if a subject did not experience the severe seizure in the baseline phase that they would not be included in the calculation of the blinded phase median seizure frequency percentage change from baseline.
Measure: Median (Inter-Quartile Range); unit: Percentage change from baseline
Arm/Group | Active Stimulation | No Stimulation
Number analyzed (Participants) | 43 | 38
Percentage change from baseline | -39.6 [-82.7 to -7.1] | -20.4 [-50.0 to 29.3]
Statistical Analysis 1: Comparison: Active Stimulation vs No Stimulation; Numbers provided indicate the percentage change from baseline in seizure frequency of each participant's most severe seizures. Negative values indicate improvement from baseline; Test type: Superiority or Other; p = 0.047, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study. The summaries below include events that occurred during the blinded phase. A summary of device related events (operative phase through Year 2) is in the safety characterization objective.
Description: Adverse events collected during the blinded phase have been included, regardless of causality.
  Because the primary purpose of this adverse event summary is to compare the randomization groups, and because the additional non-randomized subject did not have a similar follow-up schedule, the subject has not been included in these analyses.
Arm/Group | Active Stimulation | No Stimulation
Serious Adverse Events (participants affected / at risk) | 2/54 | 6/55
Other Adverse Events (participants affected / at risk) | 42/54 | 41/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (N=54) | No Stimulation (N=55)
Implant site infection (Infections and infestations) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures with secondary generalization (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (N=54) | No Stimulation (N=55)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5)
Upper respiratory infection (Infections and infestations) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 8 (8) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 0 (0)
Complex partial seizures (Nervous system disorders) | 5 (5) | 4 (4)
Memory impairment (Nervous system disorders) | 7 (7) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 2 (4) | 3 (3)
Paresthesia (Nervous system disorders) | 5 (5) | 2 (2)
Partial seizures with secondary generalization (Nervous system disorders) | 5 (5) | 3 (3)
Simple partial seizures (Nervous system disorders) | 3 (3) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 7 (8)
Anticonvulsant toxicity (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 4 (5)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)

LIMITATIONS AND CAVEATS:
No limitations leading to unreliable data were identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI allow for the sponsor to review results communications prior to public release and to embargo communications regarding trial results for a period that is less than or equal to 45 days from the time submitted to sponsor for review. The sponsor is also allowed to require changes for technical correctness and to protect confidential information, copyrightable or patentable material; and when reasonably requested, extend the embargo up to an additional 60 days.